CLINICAL TRIAL: NCT01101074
Title: A Prospective Observational Study of Safety and Effectiveness Following Administration of Adjuvanted Swine Origin A (H1N1) Pandemic Subunit Egg Derived Vaccine
Brief Title: Observational Safety and Effectiveness Study of Adjuvanted Swine Origin A (H1N1) Pandemic Subunit Egg Derived Vaccine
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V111_05
Record Dates: First submitted 2010-04-01; First posted 2010-04-09 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Influenza A (H1N1)
Keywords: Swine Flu A (H1N1) vaccine; Adjuvanted flu egg derived; Novel influenza A (H1N1): a new flu virus of swine origin
MeSH Terms: conditions — Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (6):
- 6-23 months
  Interventions: Other: This is non-intervention observational study
- 2-8 years
  Interventions: Other: This is non-intervention observational study
- 9-17 years
  Interventions: Other: This is non-intervention observational study
- 18-44 years
  Interventions: Other: This is non-intervention observational study
- 45-60 years
  Interventions: Other: This is non-intervention observational study
- >60 years
  Interventions: Other: This is non-intervention observational study

INTERVENTIONS:
Other: This is non-intervention observational study — This is non-intervention observational study

SUMMARY:
This observational study will evaluate the safety and effectiveness following administration of adjuvanted Swine Origin A (H1N1) Pandemic Subunit Egg Derived Vaccine through both an ad hoc active monitoring system and a passive surveillance of hospitalization in a large cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects resident in Emilia-Romagna and either registered with the AUSL of Reggio Emilia, Bologna, Modena and Parma or working in the province of Reggio Emilia, Bologna, Modena and Parma included in the target groups described in the Study Protocol vaccination with H1N1sw vaccine Focetria is recommended - according to the national pandemic plan adopted at the local level - will be eligible for enrolment.

Exclusion Criteria:

* Subjects already vaccinated with another pandemic vaccine or with known contraindications to Focetria, will be excluded from this study.
* Patients institutionalized in Hospital, Nursing Homes, Rehabilitation Centers, as well as home-cared patients, will also be excluded.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Population of children, adolescents, adults and elderly
Sampling Method: Non-Probability Sample
Enrollment: 135469 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety of Flu Egg Derived Adjuvanted Swine Origin A(H1N1) Pandemic Subunit Vaccine by estimating the incidence of reported Adverse Events, Serious Adverse Events or Adverse Events of Special Interest in a cohort of actively monitored vaccinated subjects | Within 3 weeks and 6 weeks after vaccine administration

SECONDARY OUTCOMES:
The occurrence of hospitalization within 6 weeks and 2 years after vaccination in a cohort of subjects vaccinated sw unvaccinated subjects, with Flu Egg Derived Adjuvanted Swine Origin A (H1N1) Pandemic Subunit Vaccine | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Emilia Romagna, Italy

REFERENCES:
- [Derived] Moro ML, Nobilio L, Voci C, Di Mario S, Candela S, Magrini N; SaFoH1N1 working group. A population based cohort study to assess the safety of pandemic influenza vaccine Focetria in Emilia-Romagna region, Italy - part two. Vaccine. 2013 Feb 27;31(10):1438-46. doi: 10.1016/j.vaccine.2012.07.090. Epub 2012 Aug 10. PMID 22885015
- [Derived] Candela S, Pergolizzi S, Ragni P, Cavuto S, Nobilio L, Di Mario S, Dragosevic V, Groth N, Magrini N; SaFoH1N1 working group. An early (3-6 weeks) active surveillance study to assess the safety of pandemic influenza vaccine Focetria in a province of Emilia-Romagna region, Italy - part one. Vaccine. 2013 Feb 27;31(10):1431-7. doi: 10.1016/j.vaccine.2012.06.030. Epub 2012 Jul 2. PMID 22766247